CLINICAL TRIAL: NCT05233813
Title: A Pilot Study of Testing the Multilevel Active Body and Mind (ABM) Intervention for Older Adults
Brief Title: Active Body and Mind Intervention for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Weiyun Chen, Associate Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00158279
Record Dates: First submitted 2022-01-13; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Well Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABM intervention group (Experimental): The intervention group received three, 45-min group exercise lessons for 12 weeks. The group exercise lessons were taught by two experienced instructors.. Each participant in the intervention group received a Fitbit (Model InspireHR) activity tracker to self-monitor their daily PA, 5 days per week for 12 weeks.
  Interventions: Behavioral: Active Body and Mind
- Comparison group (No Intervention): The comparison group continued their usual activities.

INTERVENTIONS:
Behavioral: Active Body and Mind — The intervention group attended three 45-min group exercise lessons per week and wore a Fitbit activity tracker during the weekdays for 12 weeks combined with weekly feedback and personalized activity goals.
  Arms: ABM intervention group

SUMMARY:
This study aimed to examine the effectiveness and acceptability of wearable activity trackers with self-regulatory techniques for promoting physical activity (PA) in older adults. In addition, this study aimed to investigate the impact of a multicomponent PA intervention on life satisfaction, happiness, eudaimonic well-being, and depressive symptoms, reflecting different dimensions of psychological well-being, in older adults.

DETAILED DESCRIPTION:
Fifty-nine participants living in retirement communities were voluntarily assigned to a 12-week multi-component PA intervention program or an attention control group. Participants in the intervention group were asked to take three 45-min supervised group exercise lessons per week and wear wearable activity trackers during the weekdays for 12 weeks. Four components of psychological well-being were assessed at baseline and the end of the intervention including life satisfaction, happiness, eudaimonic well-being, and depressive symptoms. The intervention effect on each component of psychological well-being was analyzed using linear mixed models after controlling for potential confounders. Participants' experiences of using the wearable activity tracker were assessed after the 12-week intervention through an 8-item questionnaire and individual interviews

ELIGIBILITY:
Inclusion Criteria:

* aged 65 or older,
* able to speak and read English fluently
* able to walk for 10 feet without human assistance

Exclusion Criteria:

* conditions preventing them from doing exercises

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Baseline Depression | Baseline (the week before the intervention)
  Depression was measured using the 10-item Centre for Epidemiological Studies Depression Inventory on a 4-point Likert scale. The level of depressive symptoms was reflected by summing the responses of the ten items, with higher scores indicating greater levels of depressive symptoms.
Baseline Happiness | Baseline (the week before the intervention)
  Happiness was measured using the 4-item Subjective Happiness Scale on a 7-point Likert scale. The mean score of all items was calculated to indicate the level of happiness with higher scores indicating greater happiness.
Baseline Life Satisfaction | Baseline (the week before the intervention)
  Life satisfaction was measured using the 5-item Satisfaction With Life Scale on a 7-point Likert scale. The sum of all items provides a composite score, with higher scores representing higher levels of life satisfaction.
Baseline Eudaimonic Well-Being | Baseline (the week before the intervention)
  Eudaimonic well-being was assessed using the 18-item Psychological Well-Being Scale on a 7-point Likert scale. An overall score was computed by averaging the scores of all items. Higher scores indicate higher levels of eudaimonic well-being.
Posttest Depression | Post-intervention test (the week after the intervention)
  Depression was measured using the 10-item Centre for Epidemiological Studies Depression Inventory on a 4-point Likert scale. The level of depressive symptoms was reflected by summing the responses of the ten items, with higher scores indicating greater levels of depressive symptoms.
Posttest Happiness | Post-intervention test (the week after the intervention)
  Happiness was measured using the 4-item Subjective Happiness Scale on a 7-point Likert scale. The mean score of all items was calculated to indicate the level of happiness with higher scores indicating greater happiness.
Posttest Life Satisfaction | Post-intervention test (the week after the intervention)
  Life satisfaction was measured using the 5-item Satisfaction With Life Scale on a 7-point Likert scale. The sum of all items provides a composite score, with higher scores representing higher levels of life satisfaction.
Posttest Eudaimonic Well-Being | Post-intervention test (the week after the intervention)
  Eudaimonic well-being was assessed using the 18-item Psychological Well-Being Scale on a 7-point Likert scale. An overall score was computed by averaging the scores of all items. Higher scores indicate higher levels of eudaimonic well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Weiyun Chen, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Z, Giordani B, Margulis A, Chen W. Efficacy and acceptability of using wearable activity trackers in older adults living in retirement communities: a mixed method study. BMC Geriatr. 2022 Mar 21;22(1):231. doi: 10.1186/s12877-022-02931-w. PMID 35313819